CLINICAL TRIAL: NCT05935306
Title: Effect of Photobiomodulation to Reduce Post-operative Pain After Endodontic Surgery: a Randomized Controlled Clinical Trial
Brief Title: Effect of Photobiomodulation to Reduce Post-operative Pain After Endodontic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Clinical Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pain after endodontic surgery
Record Dates: First submitted 2023-06-18; First posted 2023-07-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Photobiomodulation; Endodontic Disease; Pain; Inflammation; Surgery
MeSH Terms: conditions — Dental Pulp Diseases; Pain; Inflammation | interventions — Ibuprofen; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This randomized, controlled, double-blind superiority clinical trial meets the criteria for designing a clinical trial in accordance with the SPIRIT Statement. It was accepted by Research Ethics Committee (CEP) of the Catholic University of Uruguay
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Thus for the participant does not identify the group to which he belongs, the device activation sound (beep) will be recorded and it will turn on at the time of application.. Immediately after finishing the suture, the investigator in charge of applying the FBM will remove and open 1 envelope (without changing the numerical sequence of the other envelopes) and perform the indicated procedure or its simulation. Only this researcher will know the nature of the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1- Control group (Active Comparator): Conventional treatment + FBM simulation (n = 17 patients): All participants will undergo the same conventional surgical procedure. Patients will receive the FBM simulation and will be treated identically to the G2 group. The person responsible for applying the FBM will simulate the radiation by placing the devices in the same places described for the FBM group, however, the equipment will remain turned off. Thus for the participant does not identify the group to which he belongs, the device activation sound (beep) will be recorded and it will turn on at the time of application.
  Interventions: Drug: Ibuprofen; Other: Photobiomodulation simulation
- G2- Intervention group (Experimental): Conventional treatment with placebo ibuprofen + FBM (n = 17) All participants will undergo the same surgical procedure. Patients will receive FBM (Table 1) and will be treated identically to the G2 group.
  The irradiated region will be on the lesion at 4 equidistant points on the vertex of a flat square 1 cm away. A dot will be irradiated in the middle of the square (Figure 1). Placebo ibuprofen will be manipulated.
  Interventions: Device: Photobiomodulation; Other: Ibuprofen simulation

INTERVENTIONS:
Drug: Ibuprofen — All participants will undergo the same conventional surgical procedure. Patients will receive the FBM simulation and will be treated identically to the G2 group.
  Other Names: antinflamatory
  Arms: G1- Control group
Other: Photobiomodulation simulation — The person responsible for applying the FBM will simulate the radiation by placing the devices in the same places described for the FBM group, however, the equipment will remain turned off.
  Arms: G1- Control group
Device: Photobiomodulation — . Patients will receive FBM and will be treated identically to the G2 group. The irradiated region will be on the lesion at 4 equidistant points on the vertex of a flat square 1 cm away.
  Arms: G2- Intervention group
Other: Ibuprofen simulation — Placebo ibuprofen will be manipulated by pharmacy (Matias Gonzalez)
  Other Names: antinflamatory placebo
  Arms: G2- Intervention group

SUMMARY:
The objective of this study will be to evaluate if photobiomodulation (FBM) can reduce postoperative pain in patients who will undergo endodontic surgery. For this randomized, controlled and double-blind clinical study, 34 patients without comorbidities who need endodontic surgery in the upper jaw (15 to 25 teeth) will be recruited. They will be randomly divided into an experimental group (n = 17) photobiomodulation (808nm, 100 mW, and 4J/cm2 with 5 points per vestibular). Applications will be made in the immediate postoperative period and 24 hours after surgery. Control group (n = 17) a FBM simulation will be performed in the same way as in the experimental group. In this group, the required analgesia will be administered within the standard with ibuprofen. Both groups will perform the necessary conventional procedures considered the gold standard in the literature. Both the patient and the evaluator will be blinded to the intervention performed. The primary outcome variable of the study will be postoperative pain, which will be assessed using the visual analog scale at all postoperative control visits (baseline, 24 hours and 7 days). As for the secondary outcome variables, the amount of systemic medication received according to the patient's need (will be provided by the investigator).. Radiographic images will be obtained after 1 and 2 months for evaluation of the repair (dimensions of the lesion, radiopacity). These radiographs will be taken digitally with the positioners implemented. Edema, ecchymosis, and evaluation of soft tissues in the anterior portion of the intra and extra-oral maxilla will also be evaluated. In addition, a digital thermometer. These parameters will be evaluated 24 hours and 7 days after the intervention. The X-rays will be taken in the 1st and 3rd month respectively.

DETAILED DESCRIPTION:
Photobiomodulation (FBM) has shown favorable results in the postoperative period of endodontic surgery, however, up to now, the level of evidence in this procedure is low. The objective of this study will be to evaluate if photobiomodulation (FBM) can reduce postoperative pain in patients who will undergo endodontic surgery. For this randomized, controlled, and double-blind clinical study, 34 Uruguayan participants of both sexes who previously consulted at the Clínica Universitaria de la Salud, with a diagnosis of periodontitis with an apical lesion less than 10mm with or without a fistula, diagnosed clinically and radiographically, in the upper maxillary region (from 15 to 25) will be recruited. Participants included in the study must have periapical lesions who have already undergone endodontic treatment (lesions smaller than 10mm in their greatest diameter - Metin et al., 2018, single and chronic lesions), no comorbidities, age from 18 to 70 years, both genders, healthy permanent teeth with good hygiene. Participants will be excluded if they are taking drugs that affect bone metabolism and the inflammatory process (for example corticosteroids, bisphosphonates), Smokers, pregnant or lactating women, if used anti-inflammatory drugs in the last 3 months before surgery, who do not follow the guidelines or have an injury in the acute phase (pain, edema, exudate). They will be randomly divided into an experimental group (n = 17) photobiomodulation (808nm, 100 mW, and 4J/cm2 with 5 points per vestibular). Applications will be made in the immediate postoperative period and 24 hours after surgery. Control group (n = 17) FBM simulation will be performed in the same way as in the experimental group. In this group, the required analgesia will be administered within the standard with ibuprofen. Both groups will perform the necessary conventional procedures considered the gold standard in the literature. Both the patient and the evaluator will be blinded to the intervention performed. The primary outcome variable of the study will be postoperative pain, which will be assessed using the visual analog scale at all postoperative control visits (baseline, 24 hours, and 7 days). As for the secondary outcome variables, the amount of systemic medication received according to the patient's need (will be provided by the investigator). Radiographic images will be obtained after 1 and 3 months for evaluation of the repair (dimensions of the lesion, radiopacity). These radiographs will be taken digitally with the positioners implemented. Edema, ecchymosis, and evaluation of soft tissues in the anterior portion of the intra and extra-oral maxilla will also be evaluated. In addition, the temperature with a digital thermometer. These parameters will be evaluated 24 hours and 7 days after the intervention. The X-rays will be taken in the 1st and 3rd months, respectively. Once all the data have been collected, their normality will be tested, and the one-way ANOVA test and the complementary Tukey test will be carried out. Data will be presented as mean ± standard deviation (SD) and the accepted p-value will be <0.0

ELIGIBILITY:
Inclusion Criteria

:• Patients with periapical lesions who have already undergone endodontic treatment (lesions smaller than 10mm in their greatest diameter - Metin et al., 2018, single and chronic lesions)

* Patients with not comorbidities,
* Age from 18 to 70 years,
* Both genders,
* Healthy permanent teeth with good hygiene.

Exclusion Criteria:

* Who are taking drugs that affect bone metabolism and the inflammatory process (for example: corticosteroids, bisphosphonates),
* Smokers, pregnant or lactating women,
* Who used anti-inflammatory drugs in the last 3 months before surgery.
* Who for any reason interrupted the evolution of the treatment for not attending joint appointments.
* Patients who do not follow the guidelines or have an injury in the acute phase (pain, edema, exudate)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain in postoperative period - baseline | Baseline (Before the intervention)
  The primary outcome was Pain in the postoperative period, assessed using a 10 cm Visual Analogue Scale (VAS), where 0 represented "no pain" and 10 represented "worst pain imaginable." The main analysis focused on the change in pain intensity at 24 hours postoperatively compared to baseline (immediate postoperative period), as this time point is considered the most clinically relevant for evaluating the effectiveness of photobiomodulation in the management of acute postoperative pain.
Pain in postoperative period - 24 hours after treatment | 24 hours after treatment
  The primary outcome was Pain in the postoperative period, assessed using a 10 cm Visual Analogue Scale (VAS), where 0 represented "no pain" and 10 represented "worst pain imaginable." The main analysis focused on the change in pain intensity at 24 hours postoperatively compared to baseline (immediate postoperative period), as this time point is considered the most clinically relevant for evaluating the effectiveness of photobiomodulation in the management of acute postoperative pain.

SECONDARY OUTCOMES:
Pain in postoperative period - 7 days after treatment | 7th days after treatment
  Pain will also be assessed on the 7th day after surgery; however, this is defined as a secondary outcome, since other postoperative parameters-such as edema, ecchymosis, and soft tissue condition-will be evaluated at this time. Based on the literature, we do not expect significant pain at this later stage
Quantity of analgesics taken in the specific periods - baseline | Baseline (Before the intervention)
  The number of analgesics taken at the baseline will be recorded. Paracetamol will be the sole analgesic administered to the patients and recommended for use solely in cases of pain after surgery.
Quantity of analgesics taken in the specific periods - 24 hours after treatment | 24 hours after treatment
  The number of analgesics taken in the first 24 hours following surgery will be recorded. Paracetamol will be the sole analgesic administered to the patients and recommended for usage solely in cases of pain.
Quantity of analgesics taken in the specific periods - 7 days after treatment | 7 days after treatment
  The number of analgesics taken in the seven days following surgery will be recorded. Paracetamol will be the sole analgesic administered to the patients and recommended for usage solely in cases of pain.
Edema - baseline | Baseline (Before the intervention)
  A scale will be used to quantify the extent of edema. This scale has scores ranging from 0 to 3: 0 = no edema, 1 = intraoral edema, 2 = extraoral edema, and 3 = diffuse edema. This outcome will be measured at baseline, 24 hours, and seven days after surgery.
Edema - 24 hours after treatment | 24 hours after treatment
  A scale will be used to quantify the extent of edema. This scale has scores ranging from 0 to 3: 0 = no edema, 1 = intraoral edema, 2 = extraoral edema, and 3 = diffuse edema. This outcome will be measured at baseline, 24 hours, and seven days after surgery.
Edema - 7 days after treatment | 7 days after treatment
  A scale will be used to quantify the extent of edema. This scale has scores ranging from 0 to 3: 0 = no edema, 1 = intraoral edema, 2 = extraoral edema, and 3 = diffuse edema. This outcome will be measured at baseline, 24 hours, and seven days after surgery.
Ecchymosis - baseline | Baseline (Before the intervention)
  Ecchymosis refers to bleeding in the subcutaneous tissue caused by the rupture of one or more capillaries, often resulting from surgical trauma and characterized by a diameter greater than 1 cm. The assessment scale for ecchymosis is defined as follows: 0 = no color change, 1 = spot smaller than 4 cm in diameter, 2 = spot between 4 and 10 cm in diameter, 3 = spot larger than 10 cm in diameter.
Ecchymosis - 24 hours after treatment | 24 hours after treatment
  Ecchymosis refers to bleeding in the subcutaneous tissue caused by the rupture of one or more capillaries, often resulting from surgical trauma and characterized by a diameter greater than 1 cm. The assessment scale for ecchymosis is defined as follows: 0 = no color change, 1 = spot smaller than 4 cm in diameter, 2 = spot between 4 and 10 cm in diameter, 3 = spot larger than 10 cm in diameter.
Ecchymosis -7 days after treatment | 7 days after treatment
  Ecchymosis refers to bleeding in the subcutaneous tissue caused by the rupture of one or more capillaries, often resulting from surgical trauma and characterized by a diameter greater than 1 cm. The assessment scale for ecchymosis is defined as follows: 0 = no color change, 1 = spot smaller than 4 cm in diameter, 2 = spot between 4 and 10 cm in diameter, 3 = spot larger than 10 cm in diameter.
Soft tissue healing - baseline | Baseline (Before the intervention)
  Score 1: No opening along the incision line, no drainage (pus or exudate), no inflammation, and no pain. Score 2: No opening along the incision line, no drainage, mild swelling, and mild pain. Score 3: No opening along the incision line, active drainage, advanced inflammation, and moderate to severe pain. Score 4: Opening along the incision line, active drainage, advanced inflammation, and persistent pain.
Soft tissue healing - 24 hours after treatment | 24 hours after treatment
  Score 1: No opening along the incision line, no drainage (pus or exudate), no inflammation, and no pain. Score 2: No opening along the incision line, no drainage, mild swelling, and mild pain. Score 3: No opening along the incision line, active drainage, advanced inflammation, and moderate to severe pain. Score 4: Opening along the incision line, active drainage, advanced inflammation, and persistent pain.
Soft tissue healing -7 days after treatment | 7 days after treatment
  Score 1: No opening along the incision line, no drainage (pus or exudate), no inflammation, and no pain. Score 2: No opening along the incision line, no drainage, mild swelling, and mild pain. Score 3: No opening along the incision line, active drainage, advanced inflammation, and moderate to severe pain. Score 4: Opening along the incision line, active drainage, advanced inflammation, and persistent pain.
Bone consolidation - baseline | Baseline (Before the intervention)
  Bone consolidation will be assessed using periapical radiography to investigate two-dimensional changes in the bone defects. Consistent with the same equipment and employing the parallelism technique, periapical radiographs will be taken in the immediate preoperative period for comparative analysis with those taken at one and three months. The area of the defect will be determined by multiplying the longest mesiodistal and superoinferior diameters visible on the radiographs. On all radiographs, the longest diameter of the lesion will be measured. The periapical index will be determined, with the following interpretation: 0 = no lesion, 1 = periapical radiolucency with a diameter of 0.5 to 1 mm, 2 = periapical radiolucency with a diameter of 1.1 to 2 mm, 3 = periapical radiolucency with a diameter of 2.1 to 4 mm, 4 = periapical radiolucency with a diameter of 4.1 to 8 mm, and 5 = periapical radiolucency greater than 8.1 mm in diameter.
Bone consolidation - 1 month | 1 month
  Bone consolidation will be assessed using periapical radiography to investigate two-dimensional changes in the bone defects. Consistent with the same equipment and employing the parallelism technique, periapical radiographs will be taken in the immediate preoperative period for comparative analysis with those taken at one and three months. The area of the defect will be determined by multiplying the longest mesiodistal and superoinferior diameters visible on the radiographs. On all radiographs, the longest diameter of the lesion will be measured. The periapical index will be determined, with the following interpretation: 0 = no lesion, 1 = periapical radiolucency with a diameter of 0.5 to 1 mm, 2 = periapical radiolucency with a diameter of 1.1 to 2 mm, 3 = periapical radiolucency with a diameter of 2.1 to 4 mm, 4 = periapical radiolucency with a diameter of 4.1 to 8 mm, and 5 = periapical radiolucency greater than 8.1 mm in diameter.
Bone consolidation - 3 months | 3 months
  Bone consolidation will be assessed using periapical radiography to investigate two-dimensional changes in the bone defects. Consistent with the same equipment and employing the parallelism technique, periapical radiographs will be taken in the immediate preoperative period for comparative analysis with those taken at one and three months. The area of the defect will be determined by multiplying the longest mesiodistal and superoinferior diameters visible on the radiographs. On all radiographs, the longest diameter of the lesion will be measured. The periapical index will be determined, with the following interpretation: 0 = no lesion, 1 = periapical radiolucency with a diameter of 0.5 to 1 mm, 2 = periapical radiolucency with a diameter of 1.1 to 2 mm, 3 = periapical radiolucency with a diameter of 2.1 to 4 mm, 4 = periapical radiolucency with a diameter of 4.1 to 8 mm, and 5 = periapical radiolucency greater than 8.1 mm in diameter.
Local temperature - baseline | Baseline (Before the intervention)
  Temperature will be measured in degrees Celsius and compared to the baseline temperature
Local temperature - 24 hours after treatment | 24 hours after treatment
  Temperature will be measured in degrees Celsius and compared to the baseline temperature
Local temperature - 7 days after treatment | 7 days after treatment
  Temperature will be measured in degrees Celsius and compared to the baseline temperature
Sistemic temperature - baseline | Baseline (Before the intervention)
  Temperature will be measured in degrees Celsius and compared to the baseline temperature in the glabela
Sistemic temperature - 24 hours after treatment | 24 hours after treatment
  Temperature will be measured in degrees Celsius and compared to the baseline temperature in the glabela
Sistemic temperature - 7 days after treatment | 7 days after treatment
  Temperature will be measured in degrees Celsius and compared to the baseline temperature in the glabela

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Catolica do Uruguay, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: Study Protocol
Time Frame: The data will be made available upon reasonable request after the completion of the study, expected in December 2025, and will remain available for at least five years.
Access Criteria: Access to the data will be granted upon reasonable request to the corresponding author. There will be no restrictions on access, provided that the data are appropriately cited and used in accordance with ethical guidelines.
URL: https://osf.io/

REFERENCES:
- [Derived] Cirisola RWC, Moya LEP, Olazabal MVG, Wagmann DAA, Suarez GP, Wince C, Bruno MLH, Salaberry DR, Sobral APT, Longo PL, Motta LJ, Bussadori SK, Duran CCG, Fernandes KPS, Mesquita-Ferrari RA, Horliana ACRT. Photobiomodulation for postoperative pain relief following conventional periapical surgery: a randomised controlled study protocol. BMJ Open. 2025 Nov 11;15(11):e089986. doi: 10.1136/bmjopen-2024-089986. PMID 41218940